CLINICAL TRIAL: NCT02375737
Title: Evaluating CVD Medication Adherence Program in Low SES
Acronym: CVDMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: PhRMA Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00054572
Record Dates: First submitted 2015-01-16; First posted 2015-03-03 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Disease; Hypertension; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus | interventions — American Recovery and Reinvestment Act

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- m-health (Experimental): Patients will receive text message, emails, and monthly phone calls
  Interventions: Behavioral: m-health

INTERVENTIONS:
Behavioral: m-health — Patients will receive e-reminders via text message and email. A message library that allows us to disseminate constant and reliable information has been created. Messages will contain not only medication reminders, but information about issues related to self-management and medication adherence for CVD risk including messages on side-effects, risks/benefits of medication treatment, and barriers to medication adherence. In addition to these messages, patients will also receive tailored information via telephone by trained research staff.

SUMMARY:
The investigators propose to evaluate the implementation of an efficacious medication adherence program in a group at high risk for CVD. The program involves patients receiving/responding to e-reminders to take CVD medications via patient-selected technology [mobile/web-based applications, short message service (SMS; text messaging), interactive voice response (IVR), or e-mail] supported by a tailored, monthly, self-management program administered by either research staff or a case manager staff member from the Duke Outpatient Clinic via the telephone. This is a hybrid type II implementation science study.

DETAILED DESCRIPTION:
The investigators propose to evaluate the implementation of a medication adherence program among patients who attend Duke Outpatient Clinic (DOC). It is anticipated that, among the providers' patient panels, at least 100 and up to 300 with CVD risk and poor CVD medication adherence (<0.08 medication possession ratio) will consent to the program.

Using procedures from the investigators previous studies, the investigators will identify potential patients from the EHR, and will identify a pool of potential patients using electronic health records, with the goal of administering the program to at least 100 patients. Patients will be mailed letters, signed by their own provider or medical director of DOC, requesting their participation in the programs. The RA will contact patients via telephone to explain the study, screen for eligibility, and determine what mode of administration individuals prefer to receive the program (SMS, IVR, or email).

The primary outcome will be that the effectiveness/impact of the proposed adherence program will be a 10% improvement in MPR and CVD outcomes (anticipate reducing SBP by 5 mmHg, Hgb a1c by 0.5%, LDL-C by 20 mg/dl).

ELIGIBILITY:
Inclusion Criteria:

1. Medicaid recipient (preferred); however the investigators will include those patients with other types of insurance or those who are uninsured
2. Enrolled in Duke Outpatient Clinic for at least one year
3. Outpatient diagnostic code for hypertension and/or hypercholesterolemia and/or diabetes
4. Poorly controlled BP levels (>140/90) and/or LDL-C (>130mg/dl) and/or HbA1c of >8 within last 6 months

Exclusion Criteria:

1. No access to cell phone
2. Not proficient in English
3. Nursing home/long-term care facility resident or receiving home health care
4. Impaired hearing/ speech/ vision
5. Participating in another trial (pharmaceutical or behavioral)
6. Planning to leave the area in the next 12 months
7. Pregnancy (or planning)
8. Diagnosis of life-threatening disease with death probable within 1 year
9. Active Diagnosis of psychosis or dementia (has been hospitalized in the last 30 days)
10. Diagnosis of ESRD

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Adherence to the program's intervention | 6 months
  It is measured as the proportion of technology or interventionist contacts responded to by a patient out of those received over the course of the intervention period. This will be summarized descriptively by type of contact (technology vs. interventionist call) and subdivided by technology (SMS, email).

SECONDARY OUTCOMES:
Clinical effectiveness/impact of the program to pill refill adherence | 6 months
  This will be measured by pulling pill refill records of those patients who are enrolled. The investigators anticipate an improvement of 10% on pill refill adherence.
Clinical effectiveness/impact on BP | 6 months
  This will be measured by assessing systolic BP values. The investigators anticipate reducing SBP by 5 mmHg.
Clinical effectiveness/impact on A1C | 6 months
  This will be measured by assessing A1C values. The investigators anticipate reducing Hgb A1c by 0.5%.
Clinical effectiveness/impact on cholesterol | 6 months
  This will be measured by assessing LDL-C levels in patients. The goal is to reduce LDL-C levels by 20 mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Hayden Bosworth, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System Clinic, Durham, North Carolina, United States